CLINICAL TRIAL: NCT07008768
Title: Visual Outcome After Implantation of Three Different Presbyopia-correcting IOLs and Monofocal IOL
Brief Title: The Purpose is to Evaluate Visual Acuity for Distance, Intermediate and Near and Additionally Contrast Sensitivity at 25% and 10% of Illumination After Implantation of Trifocal IOL, Extended Range of Vision IOL, Bifocal IOL With Low Addition and Monofocal IOL
Acronym: IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Eye Hospital Svjetlost (Other)
Responsible Party: Principal Investigator, Mateja Jagic, MD, Principal Investigator, University Eye Hospital Svjetlost
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KS001-2018
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cataract; Presbyopia Correction; Visual Acuity
Keywords: cataract; presbyopia; visual acuity; multifocal intraocular lens
MeSH Terms: conditions — Cataract; Presbyopia | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 - TRIFOCAL IOL (Experimental): The total number of patients who underwent cataract surgery or refractive lens exchange surgery with trifocal IOL implantation was thirty of the mean (±sd; range) age 57.23 (±6.1, 45-69).
  Interventions: Procedure: Cataract surgery and refractive lens exchange surgery; Device: TRIFOCAL IOL
- Group 2 - EROV (Experimental): The total number of patients who underwent cataract surgery or refractive lens exchange surgery with extended range of vision IOL implantation was thirty-five of the mean (±sd; range) age 59.12 (±5.4, 45-71).
  Interventions: Procedure: Cataract surgery and refractive lens exchange surgery; Device: EROV IOL
- Group 3 - BIFOCAL IOL (Experimental): The total number of patients who underwent cataract surgery or refractive lens exchange surgery with bifocal IOL with low addition implantation was thirty-four of the mean (±sd; range) age 59.94 (±9.1, 45-71).
  Interventions: Procedure: Cataract surgery and refractive lens exchange surgery; Device: BIFOCAL IOL
- Group 4 - MONOFOCAL IOL (Active Comparator): The total number of patients who underwent cataract surgery or refractive lens exchange surgery with monofocal IOL implantation was thirty-two of the mean (±sd; range) age 61.33 (±8.7, 45-74), were recruited as controls.
  Interventions: Procedure: Cataract surgery and refractive lens exchange surgery; Device: MONOFOCAL IOL

INTERVENTIONS:
Procedure: Cataract surgery and refractive lens exchange surgery — Cataract surgery or refractive lens exchange surgery was performed with standard phacoemulsification procedure using micro coaxial surgical technique. After superior clear corneal incision, anterior capsulorexis and lens phacoemulsification, the IOL was implanted into the capsular bag using an injector in all cases. Ophthalmic Viscosurgical Device (OVD) was completely removed by irrigation and aspiration. All incisions were self-closing.
Device: TRIFOCAL IOL — 1-piece aspheric hydrophobic presbyopia-correcting intraocular lens, trifocal
  Arms: Group 1 - TRIFOCAL IOL
Device: EROV IOL — 1-piece aspheric hydrophobic presbyopia-correcting intraocular lens, extended range of vision (EROV)
  Arms: Group 2 - EROV
Device: BIFOCAL IOL — 1-piece aspheric hydrophobic presbyopia-correcting intraocular lens, bifocal with low addition
  Arms: Group 3 - BIFOCAL IOL
Device: MONOFOCAL IOL — Control lens: 1-piece aspheric hydrophobic monofocal aspheric IOL
  Arms: Group 4 - MONOFOCAL IOL

SUMMARY:
The objective of this study was to evaluate the effect of intraocular lens (IOL) selection on visual acuity and refractive outcomes, to assess the impact of IOL type on postoperative contrast sensitivity, and to investigate whether IOL choice influences the induction and dynamics of higher-order ocular aberrations following cataract surgery/refractive lens exchange surgery in hyperopic patients.

DETAILED DESCRIPTION:
A prospective randomized interventional clinical study was conducted in its entirety at the Department of Refractive Surgery, University Eye Hospital Svjetlost, Zagreb, Croatia. Participant enrolment occurred between January 1, 2018, and October 31, 2020. Each participant was followed prospectively for a period of 12 months.

The study was designed to include 4 groups, each comprising 50 participants. Eligible participants were those aged 45 years or older and present with hyperopia ranging from +0.50 dioptres (D) to +5.00 D, and astigmatism of up to +1.00 D. Participants with refractive errors must exhibit a best-corrected visual acuity (BCVA) of ≥0.05 Logarithm of the Minimum Angle of Resolution (LogMAR). For those with cataracts, inclusion requires a BCVA of ≥0.7 LogMAR, contingent upon cataract severity. Participants with BCVA <0.05 LogMAR were enrolled only after the exclusion of low vision, as confirmed by prior ophthalmological records.

All patients underwent a comprehensive preoperative ophthalmologic evaluation. This included slit-lamp bio microscopy of the anterior segment and dilated fundus examination. Uncorrected visual acuity (UCVA), best-corrected visual acuity (BCVA), as well as manifest and cycloplegic refractions were recorded. Corneal tomography was performed to assess the topography of both the anterior and posterior corneal surfaces, as well as corneal thickness. Wavefront aberrometry (Luneau Visionix L80 Wave+, Visionix, Prunay-le-Gillon, France), was conducted to evaluate higher-order aberrations. Pupil size was measured under photopic, mesopic, and scotopic conditions using a pupillometer (Peramis, CSO, Italy). Specular microscopy (Perseus specular microscope, CSO, Firenze, Italy), was employed to determine corneal endothelial cell density. Additional assessments included determination of ocular dominance, evaluation of ocular motility, and assessment of tear film stability using the Schirmer test and Tear Break-Up Time (TBUT) test. Contrast sensitivity (CS) at 10% and 25% illumination was also measured.

Phacoemulsification was performed using the Infinity Vision System (Abbott Medical Optics, WhiteStar Signature Phacoemulsification System). Surgical parameters, including phaco power, vacuum level, pulse mode, oscillation, and infusion bottle height, were adjusted according to the specific phase of the procedure. All surgeries were performed by a single experienced surgeon employing a standardized micro coaxial technique. Corneal incisions measuring 2.7 mm were created along the steepest meridian; in rare cases where intraoperative challenges were encountered, the incision was extended.

Following successful completion of anterior capsulorhexis and lens phacoemulsification, a foldable intraocular lens (IOL) was implanted into the capsular bag via the main incision using the Acrijet Blue injector (VSY Biotechnology, Amsterdam, Netherlands). Residual viscoelastic material was thoroughly removed by irrigation and aspiration. All corneal incisions were self-sealing and did not require suturing. At the conclusion of the procedure, an antibiotic drop was instilled intraocularly, and antibiotic ointment was applied to the conjunctival sac. Maxitrol eyedrops (Alcon, Fort Worth, Texas), a neomycin, polymyxin B sulphates, and dexamethasone ophthalmic suspension were prescribed for application after the surgery. At first postoperative day drops were administered every hour, then four times per days in first postoperative week, and then gradually tapered for next three weeks.

Patients underwent follow-up evaluations at 1 week, 1, 6, and 12 months postoperatively. During each examination, the anterior eye segment was thoroughly assessed and documented. Uncorrected and corrected visual acuity was measured at multiple working distances (6m, 80 cm and 35 cm). Additionally, refractive status was evaluated by quantifying spherical and cylindrical corrections. Contrast sensitivity was assessed under illumination levels of 10% and 25%, and higher-order aberrations of coma and SA (spherical aberration) were measured to determine optical quality.

Data from treated eyes were analysed. Details of visual acuities, sphere and cylinder refraction, contrast sensitivity at 10% and 25% illumination, and higher-order aberrations were recorded and stored on Excel spreadsheets (Microsoft, Redmond, WA) during the monitoring of the subjects. Descriptive statistics, including minimum and maximum values, means, standard deviations, medians, and interquartile ranges, were used for preliminary variable characterization by groups. Prior to inferential analyses, the Kolmogorov-Smirnov test was applied to assess the normality of variable distributions, which is a prerequisite for parametric tests such as ANOVA and the t-test. As the Kolmogorov-Smirnov test indicated non-normal distribution for the variables, nonparametric statistical methods were employed throughout subsequent analyses. Specifically, the Friedman test was utilized to evaluate differences across multiple measurement time points within groups. When the Friedman test revealed statistically significant differences, pairwise comparisons were conducted using the Wilcoxon signed-rank test to identify specific time points exhibiting significant changes. For comparisons between the two independent groups-patients implanted with a new generation multifocal intraocular lens and those receiving a monofocal lens implant-the Mann-Whitney U test was applied. All statistical tests were performed at a significance level of 0.05 (95% confidence interval).

ELIGIBILITY:
Inclusion Criteria:

* Age of ≥ 45 years
* Hyperopic correction ranging from +0.50 D to +5.00 D, and astigmatism of up to +1.00 D
* Best corrected visual acuity of ≥0.05 LogMAR

Exclusion Criteria:

* Previously performed eye surgical procedures or eye injuries
* Glaucoma
* Fuchs' endothelial dystrophy or other corneal diseases (corneal degeneration and dystrophy)
* Zonular weakness or subluxated lens
* Systemic autoimmune and rheumatic disease
* Insulin dependent diabetes

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Uncorrected and Corrected Visual Acuity changes for distance, intermediate, and near in all four groups during the follow up | 12 months
  To evaluate differences in uncorrected distance visual acuity (UDVA); corrected distance visual acuity (CDVA); uncorrected intermediate visual acuity (UIVA); corrected intermediate visual acuity (CIVA); uncorrected near visual acuity (UNVA), and corrected near visual acuity (CNVA) following the implantation of three types of multifocal intraocular lenses (IOLs) and one monofocal IOL (serving as the control group), the mean values of visual acuity parameters were compared across all four IOL groups at each postoperative measurement time point.
Higher-order aberration changes in all four groups during the follow up | 12 months
  The values of coma aberration were defined as the square root (Root mean square - RMS) of the sum of the squares of the coefficients Z-13 and Z13, while the amount of spherical aberration is defined as the value of the Z04 coefficient.
Contrast sensitivity changes at 25% and 10% illumination in all four groups during the follow up | 12 months
  Contrast sensitivity was measured monocularly on a computerized screen in a lighted room at 85cd/m2. Sloan letters were projected onto the screen at 0.1 LogMAR, at the illuminances of 25% and 10%. Visual acuity was recorded at logMAR where the patient was able to read all letters.

CONTACTS AND LOCATIONS:
Locations (1):
- Univestity Eye Hospital Svjetlost, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jagic M, Bohac M, Biscevic A, Suic SP, Patel S. Comparing Clinical Outcomes of Various Presbyopia-Correcting Intraocular Lenses Using a Novel Composite Method for the Analysis and Reporting of Uncorrected Distance, Intermediate, and Near Visual Acuities. Ophthalmol Ther. 2025 Nov 14. doi: 10.1007/s40123-025-01262-4. Online ahead of print. PMID 41239160